CLINICAL TRIAL: NCT01062269
Title: A Randomized Single Blind Placebo Controlled Single Research Site Bile Acid Sequestrant Acceptability (BASA) Scale Pilot Validation Study in Generally Healthy Subjects
Brief Title: A Single Research Site Bile Acid Sequestrant Acceptability (BASA) Scale Pilot Validation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Louisville Metabolic and Atherosclerosis Research Center (Other)
Collaborators: Provident Clinical Research (Other); Daiichi Sankyo (Industry)
Responsible Party: Harold Bays MD, L-MARC Research Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OO1
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: Bile acid sequestrant; Resin; Cholesterol; Diabetes mellitus; Lipids; Glucose; Bile Acid Sequestrant Acceptability Scale (BASA)validation study
MeSH Terms: conditions — Diabetes Mellitus | interventions — Cholestyramine Resin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cholestyramine 4 grams (Active Comparator)
  Interventions: Drug: Cholestyramine
- Cholestyramine 12 grams (Active Comparator)
  Interventions: Drug: Cholestyramine
- Tang (Placebo Comparator)
  Interventions: Drug: Tang

INTERVENTIONS:
Drug: Cholestyramine — Cholestyramine 4 grams one time dose
  Other Names: Questran
  Arms: Cholestyramine 4 grams
Drug: Cholestyramine — Cholestyramine 12 grams one dose, one day
  Other Names: Questran
  Arms: Cholestyramine 12 grams
Drug: Tang — Tang one dose one day
  Arms: Tang

SUMMARY:
The purpose of the research study is (1) to rate the taste, texture, appearance, and mixability of 2 different doses of orange flavored cholestyramine compared to orange flavored Tang, (2) rank the importance of the taste, texture, appearance, and mixability when rating cholestyramine and Tang to determine the accuracy and usefulness of a taste test questionnaire.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate patient acceptability of 2 doses of orange-flavored generic Questran (cholestyramine) versus orange-flavored Tang Drink Mix (a commercial powdered orange drink without cholestyramine) via 2 BASA scales. A second objective is to assess the 2 different versions of the BASA scale. One version will be unweighted with the score based upon the aggregate score of each acceptability component. A second version will be weighted based upon subjectively-reported importance of the acceptability components. The one main study objective or focus is to determine which version of a BASA scale best differentiates patient acceptability of a bile acid sequestrant (cholestyramine) versus a placebo control powder (containing no bile acid sequestrant) thereby determining which BASA scale is the best validated instrument for future studies in assessing and comparing patient acceptability of bile acid sequestrants.

ELIGIBILITY:
Inclusion Criteria:

Subjects or generally healthy volunteers are eligible for inclusion if they meet the following inclusion criteria during the Screening Period:

* Men or women 18-70 years of age
* In general good health.
* Subjects are capable of giving informed consent, or if appropriate, have an acceptable surrogate capable of giving consent on the subject's behalf.
* Subjects are willing and readily able to be contacted for post-study safety phone call assessments one to seven days after the single study visit.

Exclusion Criteria:

* Prior intolerance to bile acid sequestrants
* Women who are either pregnant, or who are not practicing any form of birth control.
* Prior gastrointestinal surgery
* History of ongoing gastrointestinal symptoms (indigestion, constipation, or diarrhea)
* History of bowel obstruction, malabsorption, or irritable bowel syndrome
* History of esophageal disease
* Current or past history of gall bladder disease
* Subjects enrolled in another experimental (interventional) protocol within the past 30 days prior to visit 1.
* Diagnosis of diabetes mellitus
* Known history of triglyceride levels > 300 mg/dl.
* History of alcohol or drug abuse within 1 year of study entry
* Alcohol intake that exceeds more than 2 units of alcohol drinks per day
* Blood donation within 8 weeks of the study or anticipation of blood donation during the study.
* Exposure to bile acid sequestrants (colesevelam HCl, cholestyramine, colestipol within 30 of visit 1).
* Any other situation in which the Investigator makes the judgment that participation in the study would not be in the best interest of the study participant, or in the best interest of providing reliable study data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold E Bays, MD, Principal Investigator — L-MARC Research Center
Locations (1):
- L-MARC Research Center, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in January 2010 and ended in February 2010. Enrollment officially closed on February 25th, 2010. All patient screening and study visits were conducted at L-MARC Research Center's clinic.
Pre-assignment Details: Enrolled subjects were required to meet all of the inclusion and none of the exclusion criteria prior to being randomized to a group assignment. Subjects were also required to undergo vital sign obtainment, a brief physical exam, and a medical history review to ensure they were generally healthy.
Groups:
- Cholestyramine 4 Grams vs 12 Grams vs Tang: Although 3 different arms are used in this study, there is only one study group. All subjects receive all 3 treatment arms on the same day, just in varying orders. Thus, the participant flow and baseline characteristics are the same for all three arms.
Period: Overall Study
Arm/Group | Cholestyramine 4 Grams vs 12 Grams vs Tang
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cholestyramine 4 Grams vs 12 Grams vs Tang
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants] — Although 3 different arms are used in this study, there is only one study group. All subjects receive all 3 treatment arms on the same day, just in varying orders. Thus, the age characteristics are the same for all three arms.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 40
    >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] — Although 3 different arms are used in this study, there is only one study group. All subjects receive all 3 treatment arms on the same day, just in varying orders. Thus, the age characteristics are the same for all three arms.
  years | 51.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Although 3 different arms are used in this study, there is only one study group. All subjects receive all 3 treatment arms on the same day, just in varying orders. Thus, the gender characteristics are the same for all three arms.
  Participants
    Female | 16
    Male | 26
Region of Enrollment [Number; unit: participants] — Although 3 different arms are used in this study, there is only one study group. All subjects receive all 3 treatment arms on the same day, just in varying orders. Thus, the regions of enrollment are the same for all three arms.
  participants
    United States | 42
Total Enrollment Numbers [Number; unit: Participants] — Although 3 different arms are used in this study, there is only one study group. All subjects receive all 3 treatment arms on the same day, just in varying orders. Thus, total enrollment number is reflective of all study subjects who participated in the trial.
  Participants | 42

OUTCOME MEASURES:

1. Primary Outcome: Patient Acceptability of Orange-flavored Generic Questran (Cholestyramine) vs. Tang (a Commercial Powdered Orange Drink) Via 2 Versions of a Bile Acid Sequestrant Acceptability (BASA) Scale.
Description: The Bile Acid Sequestrant Acceptability Scale has 4 scoring categories: taste, texture, appearance and mixability. Participants rank each category separately. The best possible score for each category is 5 and the worst possible score is 1.
Time Frame: 1 Day
Population: Only 42 total subjects were randomized and analyzed. However, all 42 subjects received all 3 treatment arms, just in varying order of administration.
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Cholestyramine 4 Grams | Cholestyramine 12 Grams | Tang
Number analyzed (Participants) | 42 | 42 | 42
Units on Scale
  Taste Score | 2.7 (0.1) | 2.5 (0.1) | 4.2 (0.1)
  Texture Score | 2.4 (0.2) | 2.0 (0.2) | 4.3 (0.2)
  Appearance Score | 2.8 (0.1) | 2.8 (0.1) | 4.1 (0.1)
  Mixability Score | 2.5 (0.1) | 2.1 (0.2) | 4.1 (0.1)
Statistical Analysis 1: Comparison: Cholestyramine 4 Grams vs Cholestyramine 12 Grams vs Tang; The BASA scale components were derived from the parameters best shown to differentiate acceptability between different BAS preparations (taste and texture),as well as other parameters useful for differentiating between different BAS preparations(appearance and mixability). The scale was then weighted based upon an "Importance of Acceptability" questionnaire regarding the individual scale components. The developed scale should reasonably allow for future comparisons of differing BAS formulations; Test type: Superiority or Other; p < 0.05, measures analysis of variance — Differences between test products were assessed by repeated measures analysis of variance. If sequence was not found to be statistically significant(p>0.05),then it was removed from the final model; Differences between test powders assessed by repeated measures analysis of variance, pairwise comparisons between treatments by Scheffe procedure

2. Secondary Outcome: Weighted vs. Unweighted BASA Scale
Description: The total aggregate scores for the complete BASA scale were calculated for Cholestyramine 4g, Cholestyramine 12g, and Tang. The total best possible score was 20 and the total worst possible score was 4. A weighted aggregate BASA scale score was also calculated for the Cholestyramine 4g, Cholestyramine 12g, and Tang. The best possible weighted score was 60 and the worst possible weighted score was 4.
Time Frame: 1 Day
Measure: Median (Standard Deviation); unit: Units on Scale
Arm/Group | Cholestyramine 4 Grams | Cholestyramine 12 Grams | Tang
Number analyzed (Participants) | 42 | 42 | 42
Units on Scale
  Total BASA Score | 10.3 (0.4) | 9.4 (0.4) | 16.7 (0.5)
  Weighted BASA Score | 24.8 (1.3) | 22.6 (1.2) | 41.3 (1.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed the informed consent to up to 7 days after the study visit.
Description: Adverse events were assessed in clinic during the study visit and through a follow-up phone call 1-7 days after the study visit.
Arm/Group | Cholestyramine 4 Grams | Cholestyramine 12 Grams | Tang
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 2/42 | 1/42 | 2/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholestyramine 4 Grams (N=42) | Cholestyramine 12 Grams (N=42) | Tang (N=42)
Belching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Loose Stool (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gas (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urge to have bowel movement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
(1)It was performed in generally healthy subjects, for whom lipid-altering medication may not be indicated.(2)The subjects' preference or dislike of the 1st or 2nd powder mixture might have influenced their ratings of the 2nd or 3rd powder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes